CLINICAL TRIAL: NCT00758771
Title: Using State-of-the-art Rheological Methods to Characterize CF Sputum and the Effects of Mucoactive Agents: A Pilot Study
Brief Title: Using Rheological Methods to Characterize Cystic Fibrosis (CF) Sputum and the Effects of Mucoactive Agents
Acronym: GIST
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-02116
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic Fibrosis: People who have been diagnosed with cystic fibrosis
- Healthy: People who do not have cystic fibrosis and who do not have any other lung conditions

SUMMARY:
The purpose of this study is to characterize the rheological properties of cystic fibrosis (CF) and healthy sputum and to examine the effects of mucoactive agents on the rheology of CF and healthy sputum. By collaborating with Genentech, the investigators (scientists at UCSF) plan to incorporate the latest scientific findings into our work to discover and develop new treatments for CF.

DETAILED DESCRIPTION:
There are two major mechanisms for mucus clearance in the airway, both of which are dependent upon optimal mucus viscosity and elasticity. These mechanisms are severely impaired in cystic fibrosis. The physical properties of sputum can be measured using rheological methods, enabling comparison between mucus in health and in disease. Therapies which enhance mucus clearance from the airway and decrease the volume of airway secretions are collectively called "mucoactive agents." Therapies which specifically disrupt innate mucus architecture by breaking intermolecular entanglements and bonds are called mucolytic agents. Mucolytic drugs can be considered in three general categories: classic mucolytics (n-acetylcysteine), peptide mucolytics (Pulmozyme®), and non-destructive mucolytics (hypertonic saline). Using state-of-the-art rheological methods, we can characterize the physical properties of CF mucus and measure the rheologic effects of mucoactive drugs more accurately and reproducibly than what has been previously done in the literature. In this way, we will determine which of the current mucoactive agents are most effective in normalizing sputum rheology in CF, and we will gain important insights about the limitations of current mucoactive drugs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy control subjects:

  * Age 18-65
  * No history of lung disease or cardiac disease
* Cystic fibrosis subjects:

  * Age 18-65
  * Diagnosis of CF - sweat chloride values > 60 mM on pilocarpine iontophoresis sweat tests and/or 2 allelic CF-producing mutations by genetic analysis

Exclusion Criteria:

* Use of recreational drugs within 1 year prior to enrollment
* Use of tobacco within 1 year prior to enrollment, or > 10 pack-year tobacco history
* Upper respiratory tract infection in the 4 weeks prior to enrollment in the study
* Current use of antihistamines to treat allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who have cystic fibrosis and those who do not have any lung disease
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Airway Clinical Research Center, San Francisco, California, United States

REFERENCES:
- See also: UCSF Airway Clinical Research Center website — http://airway.ucsf.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Cystic Fibrosis: Individuals who have been diagnosed with cystic fibrosis.
- Healthy: Individuals who do not have cystic fibrosis and who do not have any other lung conditions
Period: Overall Study
Arm/Group | Cystic Fibrosis | Healthy
Started | 18 | 20
Completed | 15 | 15
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Did not meet eligibility criteria | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cystic Fibrosis | Healthy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (12.8) | 41.9 (10.8) | 38.8 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 11 | 6 | 17
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Shear Rheology
Description: Baseline measure of sputum shear rheology
Time Frame: Cross-sectional
Measure: Mean (Standard Error); unit: Pascal
Arm/Group | Cystic Fibrosis | Healthy
Number analyzed (Participants) | 15 | 15
Pascal | 6.0 (2.0) | 1.8 (0.2)

ADVERSE EVENTS:
Arm/Group | Cystic Fibrosis | Healthy
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No